CLINICAL TRIAL: NCT06007183
Title: A Long-term Follow-up Study to Evaluate Safety and Immunogenicity of a Chikungunya Virus Virus-like Particle Vaccine (PXVX0317) in Healthy Adults and Adolescents After Either a Single or Booster Vaccination Dosing Regimen
Brief Title: Long-term Follow-up Study to Evaluate Safety and Immunogenicity of PXVX0317 Single or Booster Vaccination
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bavarian Nordic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: EBSI-CV-317-008
Record Dates: First submitted 2023-08-18; First posted 2023-08-23 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Chikungunya Virus Infection
Keywords: Chikungunya; PXVX0317; Vaccine; Immunogenicity; CHIKV VLP
MeSH Terms: conditions — Chikungunya Fever

STUDY DESIGN:
Intervention Model Description: All eligible participants in the youngest (12 to <18 years) and oldest 2 (≥65 years) age groups will be assigned to a booster at Year 3 (Group 1). All other participants will be randomized 1:1:1 to a booster at Year 3 (Group 1), 4 (Group 2), or 5 (Group 3). Prior to booster dose administration participants will be randomized 1:1 to CHIKV VLP vaccine booster or placebo booster.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants, care providers, and investigator will not be blinded for the timing of when the participant will receive the vaccine booster or placebo booster. They will be blinded to all booster treatment assignments (vaccine booster or placebo booster).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (7):
- Group 1a (Active Comparator): CHIKV VLP vaccine booster, 3 years post initial vaccination
  Interventions: Biological: CHIKV VLP vaccine booster
- Group 1b (Placebo Comparator): Placebo booster, 3 years post initial vaccination
  Interventions: Biological: Placebo booster
- Group 2a (Active Comparator): CHIKV VLP vaccine booster, 4 years post initial vaccination
  Interventions: Biological: CHIKV VLP vaccine booster
- Group 2b (Placebo Comparator): Placebo booster, 4 years post initial vaccination
  Interventions: Biological: Placebo booster
- Group 3a (Active Comparator): CHIKV VLP vaccine booster, 5 years post initial vaccination
  Interventions: Biological: CHIKV VLP vaccine booster
- Group 3b (Placebo Comparator): Placebo booster, 5 years post initial vaccination
  Interventions: Biological: Placebo booster
- Group 4 (No Intervention): Unrandomized or unboosted participants, for any reason

INTERVENTIONS:
Biological: CHIKV VLP vaccine booster — CHIKV VLP vaccine is comprised of chikungunya virus virus-like particles (CHIKV VLP) 40mg, aluminum hydroxide 2% adjuvant, and formulation buffer supplied as a single dose of 0.8 mL in a pre-filled syringe, to be administered via intramuscular (IM) injection in the deltoid muscle.
  Other Names: PXVX0317
  Arms: Group 1a; Group 2a; Group 3a
Biological: Placebo booster — Placebo is comprised of formulation buffer supplied as a single dose of 0.8 mL in a pre-filled syringe administered via IM injection in the deltoid muscle.
  Arms: Group 1b; Group 2b; Group 3b

SUMMARY:
The purpose of this phase 3 multicenter, randomized, double-blind, placebo-controlled rollover study is to evaluate the safety and long-term immunogenicity of CHIKV VLP vaccine in adult and adolescent participants and to evaluate CHIKV VLP booster vaccine induced serum neutralizing antibody (SNA) response at 3, 4, or 5 years post-initial CHIKV VLP vaccination.

DETAILED DESCRIPTION:
Primary Objectives:

* To evaluate the long-term immunogenicity of CHIKV VLP vaccine in healthy adult and adolescent participants as measured by proportion of participants maintaining an anti-CHIKV serum neutralizing antibody (SNA) titer ≥100 (seroresponse rate, also considered the presumptive seroprotection rate) at yearly intervals up to 5 years postvaccination in feeder studies EBSI-CV-317-004 (NCT05072080) and EBSI-CV-317-005 (NCT05349617).
* To assess the vaccine-induced SNA titers by a booster dose of CHIKV VLP vaccine at 3, 4, or 5 years post-initial vaccination in feeder studies EBSI-CV- 317-004 and EBSI-CV-317-005.
* To evaluate the safety and tolerability of CHIKV VLP vaccine in all participants.
* To evaluate the safety and tolerability of a booster vaccination and compare with safety and tolerability reported post-initial vaccination of CHIKV VLP vaccine under feeder studies EBSI-CV-317-004 and EBSI-CV-317-005 in healthy adults and adolescents.

Secondary Objectives:

* To evaluate the long-term immunogenicity of CHIKV VLP vaccine in healthy adult and adolescent participants as measured by anti-CHIKV SNA geometric mean titers (GMTs) at yearly intervals up to 5 years post-initial vaccination in feeder studies EBSI-CV-317-004 and EBSI-CV-317-005.
* To evaluate the immune response to a booster vaccination and compare this response to that reported post-initial vaccination of CHIKV VLP vaccine under feeder studies EBSI-CV-317-004 and EBSI-CV-317-005 in healthy adults and adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Only within the EBSI-CV-317-004 feeder study informed consent form (ICF) (and/or assent form, as applicable), the participant voluntarily signed and agreed to be contacted or did not indicate they were not to be contacted for potential screening and enrollment in a future study (ie, EBSI-CV-317-008).
* Able and willing to provide informed consent (and assent, as applicable) voluntarily signed by participant (and guardian, as applicable) for participation in this rollover study EBSI-CV-317-008, including possible receipt of a booster dose of CHIKV VLP vaccine.
* Males or females, 12 years of age or older at the time of enrollment in the feeder study.
* Received a single dose of CHIKV VLP vaccine in one of the feeder studies, EBSI-CV-317-004 or EBSI-CV-317-005.
* Demonstrated compliance to the feeder study conduct (ie, rollover participant was without protocol deviations that excluded them from immunogenicity analysis in feeder study EBSI-CV-317-004 or EBSI-CV-317-005) without discontinuation or early withdrawal.
* Generally healthy, in the opinion of the investigator, based on medical history and physical examination.

Additional inclusion criteria to be assessed at Prerandomization Visit (Visit 5), before Randomization A (Visit 6), and before Randomization B (Visit 8 for Group 2 and Visit 10 for Group 3) to determine eligibility for a booster dose of CHIKV VLP vaccine or placebo:

- Women who are either: i. Not of childbearing potential (CBP): premenarche, surgically sterile (at least six weeks postbilateral tubal ligation or bilateral total salpingectomy, bilateral oophorectomy, or hysterectomy), or postmenopausal (defined as a history of ≥12 consecutive months without menses prior to randomization in the absence of other pathologic or physiologic causes, following cessation of exogenous sex-hormonal treatment). For women who are postmenopausal, documented follicle stimulating hormone (FSH) level of ≥40 mIU/mL must be obtained. If the FSH is <40 mIU/mL, the participant must agree to use an acceptable form of contraception. or: ii. Meet all the below criteria:

* Negative serum pregnancy test at Prerandomization and Prebooster Visits
* Negative urine pregnancy test immediately prior to booster dose administration
* Use one of these acceptable methods of contraception (if women of CBP) for at least six months after booster:
* Hormonal contraceptives (eg, implants, pills, patches) initiated ≥30 days prior to booster dose administration
* Intrauterine device (IUD) inserted ≥30 days prior to booster dose administration
* Double barrier type of birth control (male condom with female diaphragm, male condom with cervical cap)
* Abstinence is acceptable only for adolescents (12-<18 years of age) who are not sexually active.

Women participants of CBP must use an acceptable method of contraception from ≥30 days prior to Randomization A or assignment to Group 1; those who are randomized to Groups 2 or 3 at year 3 can discontinue contraception until 30 days prior to booster dose administration, if desired. Women participants of CBP must use an acceptable method of contraception from ≥30 days prior to Randomization B through six-months postbooster vaccination dose (if applicable).

Note: Contraception requirements do not apply for participants in exclusively same-sex relationships and these participants should have no plans to become pregnant by any other means during the same time period as women of CBP are required to use contraception. Contraception requirements do not apply to Group 4 participants (unrandomized or unboosted).

Exclusion Criteria:

* Received placebo treatment in the feeder study.
* Measurable anti-CHIKV SNA at Day 1 in the feeder study.
* History of severe allergic reaction or anaphylaxis to any component of the investigational product (IP).
* Receipt of either an investigational or licensed CHIKV vaccine (excluding prior receipt of CHIKV VLP vaccine).
* New onset/diagnosis of any disease falling within the feeder study exclusion criteria including: i. History of any known congenital or acquired immunodeficiency that could impact response to vaccination (eg, leukemia, lymphoma, generalized malignancy, functional or anatomic asplenia, alcoholic cirrhosis) or ii. Clinically significant cardiac, pulmonary, rheumatologic, or other chronic disease, in the opinion of the investigator. This may include chronic illness requiring hospitalization during the feeder study.
* Evidence of substance abuse that, in the opinion of the investigator, could adversely impact the individual's participation or the conduct of the study.
* Any other medical condition or general reason that, in the opinion of the investigator, could adversely impact the individual's participation or the conduct of the study.
* Bavarian Nordic staff members and their families, contractors, agents, business partners, and anyone with a financial interest in the outcome of the study.

Additional exclusion criteria to be assessed at Prerandomization Visit (Visit 5), before Randomization A (Visit 6), and before Randomization B (Visit 8 for Group 2 and Visit 10 for Group 3) to determine eligibility for a booster dose of CHIKV VLP vaccine or placebo:

* Participation or planned participation in an investigational clinical trial, excluding feeder studies EBSI-CV-317-004 or EBSI-CV-317-005 (eg, vaccine, drug, medical device, or medical procedure) for the following time periods:

Group 1: 30 days prior to Randomization A or assignment to Group 1 at Visit 6 through Visit 7 Group 2: 30 days prior to Randomization A at Visit 6 until the Randomization A visit and 30 days prior to booster dose at Visit 8 through Visit 9 Group 3: 30 days prior to Randomization A at Visit 6 until the Randomization A visit and 30 days prior to booster dose at Visit 10 through EOS Visit Group 4: 30 days prior to Randomization A at Visit 6 until the Randomization A visit Note: Participation in an observational trial or follow-up phase of a trial may be allowed; however, these instances should be discussed with this study's medical monitor (MM).

* Currently breastfeeding.
* Positive laboratory evidence of current infection with human immunodeficiency virus (HIV), hepatitis C virus (HCV) or hepatitis B virus (HBV).
* Prior receipt or anticipated use of systemic immunomodulatory or immunosuppressive medications from six months prior to Prebooster Visit through 21 days after booster dose. Note: For systemic corticosteroids, use at a dose or equivalent dose of 20 mg of prednisone daily for 14 days or more within three months of Prebooster Visit through 21 days postbooster dose is exclusionary. The use of inhaled, intranasal, topical, ocular, or intraocular steroids is allowed.
* Receipt or anticipated receipt of blood or blood-derived products from 90 days prior to Prebooster Visit through 21 days postbooster dose.
* Acute disease within the last 14 days prior to booster dose (participants with an acute mild febrile illness can be considered for a deferral of vaccination two weeks after the illness has resolved and treatment has been completed).
* Receipt or anticipated receipt of any vaccine from 30 days prior to booster dose through 21 days postbooster.

Note: Participants that are ineligible or decline booster will be included in Group 4 (unrandomized or unboosted) for follow-up unless consent/assent for follow-up is withdrawn.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2023-08-30 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants maintaining a preboost anti-CHIKV SNA titer ≥100 at yearly intervals up to 5 years post-initial vaccination | 5 years post-initial vaccination in feeder study EBSI-CV-317-004 or EBSI-CV317-005 until booster
  For all groups using the immunogenicity evaluable population (IEP) the proportion of participants maintaining a preboost anti-CHIKV SNA titer ≥100 (seroresponse rate, also considered the presumptive seroprotection rate) at yearly intervals up to 5 years post-initial vaccination in one of the feeder studies; only prebooster data will be summarized.
Proportion of vaccine boosted participants with composite booster response at 21 days after booster vaccination | 21 days after booster vaccination
  For IEP participants who receive a CHIKV VLP vaccine booster (Groups 1a, 2a, and 3a), proportion of participants with a boost response is defined as a composite of:
  * ≥4-fold rise in anti-CHIKV SNA titer from prebooster to postbooster measured at 21 days after booster for participants with a prebooster titer ≥100 OR
  * Anti-CHIKV SNA titer ≥100 and ≥4-fold increase in anti-CHIKV SNA titer from prebooster to postbooster measured at 21 days after booster vaccination for participants with a prebooster titer <100.
  Note: Prebooster is the last SNA sample prior to booster dose, ideally the sample on boost day prior to booster dose administration but can be the time point prior if the boost day sample is missed or incorrectly processed.

SECONDARY OUTCOMES:
Anti-CHIKV SNA Geometric Mean Titers (GMTs) at yearly intervals | 5 years post-initial vaccination in feeder study EBSI-CV-317-004 or EBSI-CV-317-005 until booster
  For all groups using the IEP, anti-CHIKV SNA GMTs preboost at yearly intervals up to 5 years post-initial CHIKV VLP vaccination in feeder study EBSI-CV-317-004 or EBSI-CV-317-005; only prebooster data will be summarized.
Anti-CHIKV SNA GMTs at 21 days postboost | 21 days postboost for Groups 1a, 2a, and 3a
  Anti-CHIKV SNA GMTs in Groups 1a, 2a, and 3a (PXVX0317 IEP booster population), at 21 days postboost.
Anti-CHIKV SNA Geometric Mean Fold Increase (GMFI) Prebooster to Postbooster | 21 days after booster vaccination and 5 years post-initial vaccination in feeder study EBSI-CV-317-004 or EBSI-CV-317-005
  For IEP participants who receive a CHIKV VLP vaccine booster (Groups 1a, 2a, and 3a) and have a 21-day postbooster SNA titer, GMFI from prebooster anti-CHIKV SNA titer to 21 days postbooster anti-CHIKV SNA titer and at yearly intervals up to 5 years post-initial vaccination in feeder study EBSI-CV-317-004 or EBSI-CV-317-005.
Booster Response at 21 Days Relative to 21-day Response in Feeder Study EBSI-CV-317-004 or EBSI-CV-317-005 | 21 days after booster vaccination
  For IEP participants who receive a CHIKV VLP vaccine booster (Groups 1a, 2a, and 3a) and have a 21-day postboost SNA titer, GMFI from feeder study EBSI-CV-317-004 or EBSI-CV-317-005 Day 22 SNA titer to 21-day postbooster SNA titer in the rollover study.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Ajiboye, MD, Study Director — Bavarian Nordic
Locations (24):
- United States (24):
  - Alliance for Multispecialty Research, LLC, Mobile, Alabama
  - Alliance for Multispecialty Research, LLC, Tempe, Arizona
  - Optimal Research, LLC, Melbourne, Florida
  - Suncoast Research Associates, LLC, Miami, Florida
  - Synexus Clinical Research US, Inc., Chicago, Illinois
  - Optimal Research, LLC, Peoria, Illinois
  - Alliance for Multispecialty Research, LLC, Newton, Kansas
  - Alliance for Multispecialty Research, LLC, Wichita, Kansas
  - Alliance for Multispecialty Research, LLC, Lexington, Kentucky
  - Alliance for Multispecialty Research, LLC, Kansas City, Missouri
  - Wr-Crcn, Llc, Las Vegas, Nevada
  - Alliance for Multispecialty Research, LLC, Las Vegas, Nevada
  - Rochester Clinical Research, LLC, Rochester, New York
  - M3 Wake Research Inc., Raleigh, North Carolina
  - Velocity Clinical Research, Cleveland, Cleveland, Ohio
  - Lynn Institute of Norman, Norman, Oklahoma
  - Velocity Clinical Research, Medford, Medford, Oregon
  - Velocity Clinical Research, Providence, East Greenwich, Rhode Island
  - Velocity Clinical Research, Austin, Cedar Park, Texas
  - DM Clinical Research, Houston, Texas
  - BFHC Research, LLC, San Antonio, Texas
  - DM Clinical Research, Tomball, Texas
  - Velocity Clinical Research, Salt Lake City, West Jordan, Utah
  - Alliance for Multispecialty Research, LLC, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No